CLINICAL TRIAL: NCT04966585
Title: A Multicenter Randomized, Double-Blinded, Placebo-Controlled Study of Posaconazole in Genetically-Defined Patients With Active Crohn's Disease
Brief Title: Pilot Study of Posaconazole in Crohn's Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment challenges; changes in manufacturing
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Gil Melmed, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MOD03104; 1R01DK125495-01A1 (NIH)
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Crohn Disease; CARD9 S12N Risk Allele
Keywords: Crohn's; Malassezia; CARD9 S12N; Antifungal
MeSH Terms: conditions — Crohn Disease | interventions — posaconazole

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to receive posaconazole or placebo in 1:1 fashion.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Both subject and clinical staff will be masked to treatment group assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Posaconazole (Experimental): Subjects administered posaconazole (Noxafil®, Merck) 300mg twice daily for 1 day followed by 300mg daily for 12 weeks
  Interventions: Drug: Posaconazole Delayed Release Oral Tablet
- Placebo (Placebo Comparator): Subjects administered three matching placebo tablets twice daily for 1 day followed by three tablets daily for 12 weeks
  Interventions: Drug: Matching Placebo Tablet

INTERVENTIONS:
Drug: Posaconazole Delayed Release Oral Tablet — Three 100mg delayed-release tablets twice a day on the first day, then three 100mg delayed-release tablets once a day, starting on the second day. Duration of therapy will be 12 weeks.
  Other Names: Noxafil
  Arms: Posaconazole
Drug: Matching Placebo Tablet — Three matching placebo tablets twice a day on the first day, then three tablets once a day, starting on the second day. Duration of therapy will be 12 weeks.
  Arms: Placebo

SUMMARY:
This trial is designed to evaluate the effects of oral antifungal treatment with posaconazole on active Crohn's disease (CD) activity and the burden of Malassezia spp. in CD patients with the caspase recruitment domain family member 9 (CARD9) S12N risk allele. Further, this project will investigate the hypothesis that the microbial changes induced by antifungal treatment are associated with dampened downstream immune responses in those with a genetic predisposition to developing strong immune responses to Malassezia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years and older, inclusive based on the date of the screening visit.
* A diagnosis of CD with minimum disease duration of 6 months with involvement of the ileum and/or colon documented on colonoscopy
* Have an endoscopically-confirmed active Crohn's disease with active disease defined by SES-CD > 6 (>4 if ileal only), AND active symptoms of Crohn's disease (CDAI score >220)
* Homozygous for CARD9 S12N risk allele, without the protective exon 11 polymorphism
* Subjects receiving oral aminosalicylates (at a stable dose for 2 weeks prior to baseline), immunomodulators (at a stable dose for 4 weeks prior to baseline), anti-TNF, anti IL12/23, or anti-integrin therapy (at stable maintenance doses for > 8 weeks) may continue their use during the study.
* Subjects receiving oral corticosteroids may continue their use during the study provided the dose (prednisone up to 20 mg/day, budesonide up to 9 mg/day) has been stable for two weeks prior to screening.
* Have had age-appropriate and disease-duration-appropriate colon cancer screening1 without unresected dysplasia.
* Women of childbearing age, excluding those with prior bilateral tubal ligation or at least one-year post-menopause, must not be pregnant, lactating, or planning to become pregnant. They must agree to use effective contraception throughout the study period.
* Subjects must be able to provide informed consent and understand, agree with, and be able to adhere to daily diary entries, all scheduled visits, tests, procedures, and protocol in English.

Exclusion Criteria:

* Known hypersensitivity or allergy to posaconazole or other azole antifungal agents
* Concomitant medications primarily metabolized by CY3PA4 including: a) Hydroxymethylglutaryl-CoA (HMG-CoA) reductase inhibitors, primarily metabolized by CY3PA4 (increases risk of rhabdomyolysis), b) Sirolimus, c) Ergot alkaloids, d) vincristine
* Proarrhythmic conditions
* Moderate or severe renal impairment (Cr Clearance <50)
* Current diagnosis of ulcerative colitis, indeterminate colitis, ischemic colitis, infectious colitis, or microscopic colitis.
* Fulminant colitis, toxic megacolon, peritonitis, ileostomy or colostomy.
* Stool sample positive for pathogens including ova and parasites, Salmonella, Shigella, and C. difficile at screening.
* History of any clinically significant neurological, renal, hepatic, gastrointestinal, pulmonary, metabolic, cardiovascular, psychiatric, endocrine, hematological disorder or disease or any other medical condition that, in the Investigators opinion, would prevent the subject from participation in the study.
* Treatment with antibiotics, antifungal agents, probiotics, or prebiotics within two weeks of screening.
* Alcohol or drug abuse (in the opinion of the Investigator) that would interfere with compliance.
* Any other investigational therapy or treatment within four weeks of screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Endoscopic Response | Week 12
  Defined as ≥ 50% reduction from baseline in Simple Endoscopic Score for Crohn's Disease (SES-CD). The SES-CD evaluates 4 endoscopic variables: ulcer size, ulcerated surface, affected surface, and presence of narrowings. The total SES-CD is calculated as the sum of the 4 variables for the 5 bowel segments: rectum, left colon, transverse colon, right colon, and ileum. Scores range from 0 to 60, with higher scores indicating more severe disease.

SECONDARY OUTCOMES:
Induction of Clinical Remission | Week 12
  Defined as Patient-Reported Outcome (PRO2) abdominal pain score ≤1 AND stool frequency ≤3, and Crohn's Disease Activity Index (CDAI) (<150).
  PRO2 is the weighted average of the 2 variables of frequency of liquid or very soft stool and abdominal pain, based on 7-day participant diary data. The PRO2 score has a minimum score of 0 and has no upper bound, with a higher score indicating more frequent stools and more severe abdominal pain.
  The CDAI is a weighted, composite index of 8 disease variables (stool frequency, severity of abdominal pain, degree of general well-being, presence or absence of extra-intestinal manifestations or fistula, use or non-use of antidiarrheal agents, presence or absence of an abdominal mass, hematocrit, and body weight). Scores range from approximately 0 to 600, with a higher score indicating more-severe disease activity.
Incidence of adverse events | Week 12
Change in amount of concomitant medications | Week 12
Proportion of subjects in endoscopic remission | Week 12
  Defined as a Simple Endoscopic Score for Crohn's Disease (SES-CD) score of ≤3. The SES-CD evaluates 4 endoscopic variables: ulcer size, ulcerated surface, affected surface, and presence of narrowings. The total SES-CD is calculated as the sum of the 4 variables for the 5 bowel segments: rectum, left colon, transverse colon, right colon, and ileum. Scores range from 0 to 56, with higher scores indicating more severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: Gil Y Melmed, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center (CSMC), Los Angeles, California
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT04966585/ICF_000.pdf